CLINICAL TRIAL: NCT00987597
Title: Effectiveness of a Managed Care Smoking Cessation Program in Patients With Acute Coronary Syndrome Based on Nicotine Replacement as a Treatment and a Cognitive-behavioral Approach
Brief Title: Smoking Cessation for Patients With Acute Coronary Syndrome (ACS)
Acronym: PATPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LRB0801; EUDRACT : 2008-00267712; ID RCB : 2008-A00509-46
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2013-11

CONDITIONS: Smoking; Acute Coronary Syndrome
Keywords: Smoking; nicotine replacement; psychological behaviour; Smoking > 5 cigarettes per day; Hospitalisation for acute coronary syndrome
MeSH Terms: conditions — Smoking; Acute Coronary Syndrome | interventions — Tobacco Products; Health Planning Guidelines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cognitive behavioural approach (Experimental): specific technique of cigarette exposure and nicotinic treatment adjustment
  Interventions: Behavioral: Technique of in-vivo exposure (cigarette) and mental image exposure (craving)
- usual approach (Active Comparator): recommendations and nicotinic substitutes
  Interventions: Behavioral: conventional follow-up

INTERVENTIONS:
Behavioral: Technique of in-vivo exposure (cigarette) and mental image exposure (craving) — Nicotine replacement
  Other Names: Reduce the urge to smoke; Strategies to avoid the relapse
  Arms: cognitive behavioural approach
Behavioral: conventional follow-up — nicotinic substitutes
  Other Names: recommendations
  Arms: usual approach

SUMMARY:
The aim of the present study is to assess if a personal care program of smokers hospitalised for acute coronary syndrome can change the smoking habits as compared with similar patients in conventional care program at 6 months. The program includes a cognitive-behavioural approach associated with a nicotine replacement treatment presented as an obligatory non optional treatment. Patients are men and women of less than 70 years old hospitalised for acute coronary syndrome. Major exclusion criteria is the presence of another dependence. The program includes a cognitive-behavioural approach based on the specific technique of "exposure" and the prescription of nicotine patch considered as other usual cardiologic treatments for at least 6 months. The end point is the smoking habits at 6 months classified as: no smoking confirmed by CO measurement, smoking or doubtful (declaration of no smoking by the patient but a CO level > 10 ppm). 72 patients in each group will be included in 2 majors sites.

DETAILED DESCRIPTION:
The cognitive behavioural approach group : This group will receive an inclusion visit at first, then two "cigaret exposures cessions" during hospitalisation. Thereafter-one week after he's out- the patient will come for 5 follow up visits consisting in the specific technique of cigaret exposure and nicotinic treatment adjustment. Then the last visit, at six months, will tell us if the patient is an effective non smoker or not; We'll be also collecting psychological and medical informations (such as the treatment, IMC, cardiovascular check up and psychological tests). The control group : This group is managed as "usual" : the nurse gives very rapid recommendations to the patients concerning smoking cessation. Nicotinic substitutes are proposed to the patients but the patient must find them by itself.

ELIGIBILITY:
Inclusion Criteria:

* Patients are men and women of less than 70 years old
* Hospitalised for acute coronary syndrome in cardiology Intensive Care Unit
* Active smoking >5 cigarettes/day
* Has given consent to participate in the study and haven't expressed its opposition the exploitation of data as part of the study

Exclusion Criteria:

* Presence of another dependence : alcohol abuse avowed or strongly suspected, addiction to drugs, high dose benzodiazepine dependence. clinical assessment
* Major psychiatric disorders or history. clinical assessment
* Treatment with lithium and neuroleptic. clinical assessment
* Patient whose cardiac problem could lead to hemodynamic instability during 48 h after admission.
* Patient scheduled for programmed hospitalisation within 6 months after release from hospital (>3 days long, including coronary bypass)
* Patients presenting another severe pathology requiring 6 months specific treatments. clinical assessment
* Patient which cannot understand or read French
* Patient with possible side-effect to nicotine substitute
* Patient unaffiliated to any social security regime

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The smoking habits at 6 months classified as : no smoking confirmed by CO measurement, smoking or doubtful (declaration of no smoking by the patient but a CO level > 10 ppm). | 6 month

SECONDARY OUTCOMES:
Assessment depending of age classes, sex, anxiety scale and other psychological characteristics | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Patrick HENRY, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Laurent MAGNE, Study Director — Cabinet MAGNE & GALLY; Olivia GALLY, Study Director — Cabinet MAGNE & GALLY
Locations (1):
- CHU Lariboisière, APHP, Cardiology, Paris, Île-de-France Region, France